CLINICAL TRIAL: NCT05553132
Title: Hip RECLAIM: A Phase I Safety and Feasibility Trial of REcycled CartiLage Auto/Allo IMplantation for the Treatment and Repair of Focal Hip Cartilage Defects
Brief Title: A Study of REcycled CartiLage Auto/Allo IMplantation to Treat and Repair Focal Hip Cartilage Defects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel B. F. Saris (Other)
Responsible Party: Sponsor-Investigator, Daniel B. F. Saris, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-004639
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cartilage Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CartiLage Auto/Allo IMplantation for Focal Hip Cartilage Defects (Experimental): Subject will receive the combined product of autologous cartilage cells and allogeneic AMSCs in a fibrin glue carrier.
  Interventions: Combination Product: Autologous Chondrocytes in their Pericellular Matrix (Chondrons) Coimplanted with Allogeneic Adipose-Derived Mesenchymal Stromal Cells (AMSCs) in a Fibrin Glue Carrier

INTERVENTIONS:
Combination Product: Autologous Chondrocytes in their Pericellular Matrix (Chondrons) Coimplanted with Allogeneic Adipose-Derived Mesenchymal Stromal Cells (AMSCs) in a Fibrin Glue Carrier — Cartilage cells are being used from the rim of the defect in the hip and recycled to help make new cartilage in the hip. There are not enough cartilage cells to fill the defect so cartilage cells need to be mixed with MSCs. MSCs or Mesenchymal Stem Cells are naturally occurring cells that provide growth factors and cell signals that play a role in tissue repair. MSCs can be found in bone marrow and in the fatty tissues (i.e., area under the skin of the belly or breast) of patients. Fibrin glue is a product made from the naturally occurring compounds in blood which cause clotting. This glue hardens into a gel-like substance into which cells such as cartilage cells (chondrons) and AMSCs can be placed.

SUMMARY:
The purpose of this research study it to gather information on the safety and side effects of treating cartilage defects with autologous cartilage cells mixed with allogeneic adipose-derived mesenchymal stem cells (AMSCs) in a fibrin glue.

ELIGIBILITY:
Inclusion Criteria:

* Persons of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal or barrier method or abstinence) at the time of screening. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered, and the result will be confirmed by a serum pregnancy test. Urine pregnancy tests will be performed by qualified personnel using kit. Persons becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded.
* Chronic (> 3 months), unilaterally symptomatic, ICRS Grade III or IV cartilage lesions ranging in size from 2 to 6 cm2. Patients with episodes of contralateral hip pain that is asymptomatic at the time of enrollment will be eligible for inclusion. However, patients with previous episodes of contralateral hip pain who experience a repeat episode of contralateral pain similar to their established pattern of pain during the course of the trial will not be considered as having experienced an adverse event.
* Radiographic hip OA of Tönnis Grade 1 or less, consisting of normal hip radiographs (Grade 0) or doubtful narrowing of the joint space and possible osteophytic lipping (Grade 1) as agreed upon by two study co-investigators without underlying structural hip abnormalities
* Previous 6 week or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications, or injection therapy (e.g. cortisone). An adequate trial will consist of pursuance and reasonable execution (i.e. > 80% medication or therapy compliance) of medically reasonable course of non-operative modalities with minimal to no improvements in symptoms
* If applicable, at least 3 months will have passed since the last target hip intraarticular injection prior to undergoing the RECLAIM procedure and at least 6 months will have passed between any prior arthroscopic or open hip procedures.
* Able to routinely walk without assistance (e.g. cane, walker)
* Clinically stable target hip.
* No additional surgery planned in the target hip for at least 12 months following the RECLAIM procedure
* Completed general physical and well-being evaluation with primary care provider within 12 months of enrollment
* Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including laboratory tests, diagnostic imaging, and follow-up visits and assessments
* Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure

Exclusion Criteria:

* Pregnant or nursing, or planning on becoming pregnant during the study period
* Congenital or acquired malformation of the target hip resulting in significant deformity or leading to problems with the study treatment or analysis of the results
* Significant structural deformity, including large cam lesion (alpha angle greater than 55 degrees) or moderate dysplasia (defined as lateral center edge angle less than 18 degrees).
* Injections of any kind into the target hip within 3 months prior to study enrollment
* History of intra-articular infection in the target hip
* History of superficial infection in the target hip within 6 months of study enrollment, or evidence of current superficial infection affecting the target hip
* History of falls requiring medical attention, or gait instability
* Clinically significant abnormal hematology (complete blood count with differential), blood chemistry, or urinalysis screening laboratory results. Absolute cutoffs for exclusion include hemoglobin < 11 g / dL, platelets < 110,000 platelets / mL, and an INR greater than 1.3.
* Body mass index (BMI) > 35 kg/m2
* Tönnis Grade II or greater on X-Ray.
* Taking anticoagulant medications (e.g. warfarin, heparin or clopidogrel) which may pose a clinically significant contraindication to the surgical RECLAIM procedure
* Taking herbal therapies or supplements within 4 weeks of enrollment or unwilling to avoid use of herbal therapies or supplements until study completion (includes, but not limited to chondroitin sulfate, diacerein, n-glucosamine, piascledine, and capsaicin)
* Taking non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) without a stable dosing regimen for at least 4 weeks before baseline evaluation, or anticipating not remaining on a stable dose until study completion
* On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
* Current tobacco product use, including nicotine patch or other nicotine products
* Clinically significant rheumatological or inflammatory disease of the hip or chondrocalcinosis/calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the hip associated with juxta-articular Paget's disease of the femur or pelvis, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's hip joint, villonodular synovitis, and synovial chondromatosis
* Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis
* Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension), neurologic (e.g. stroke, TIA) renal, hepatic, orthopedic (e.g. surgery on other weight bearing joints that will interfere with study, osteoporosis, acute lower body fractures), or endocrine disease (e.g. diabetes).
* Any clinically significant comorbidity affecting the patient's ability to undergo surgery
* Vascular or neurological disorder affecting the either lower limb which poses clinical significance to the safety of the operative RECLAIM procedure.
* History of cancer/malignancy with the exception of adequately treated basal cell or squamous cell carcinoma of the skin not associated with the target knee
* History of clinically significant blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy
* Participation in a study of an experimental drug or medical device within 3 months of study enrollment
* Known allergy to local anesthetics or other components of the study drug. This includes known allergy or contraindications to products of bovine origin (including aprotinin) or hypersensitivity to antibiotics, if the latter are used in the manufacturing process
* Any contraindication to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures
* Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* History of coagulopathy, including bleeding diathesis and deep venous thrombosis/pulmonary embolism.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 2 years
  Number of adverse events defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship.
Incidence of serious adverse events (SAEs) | 2 years
  Number of SAEs as defined as AEs that result in death, life threatening adverse experiences, hospitalization, new or prolonged disability/incapacity, persistent or significant congenital defect/anomaly, or other events that in the opinion of the PI may have adversely affected the rights, safety, or welfare of the subjects or others, or substantially compromised the research data.

SECONDARY OUTCOMES:
Change in pain | Baseline, 1-2 weeks, 6 weeks, 12 weeks, 24 weeks, 52 weeks, 18 months, and 24 months post-treatment
  Measured using self-reported 10 mm VAS
Change in physical function | Baseline, 1-2 weeks, 6 weeks, 12 weeks, 24 weeks, 52 weeks, 18 months, and 24 months post-treatment
  Measured using the PROMIS-CAT-Physical Function assessment with questions to evaluate self-reported physical function on a scale of 5 to 1, with higher scores indicating better outcomes.
Change in hip function | Baseline, 1-2 weeks, 6 weeks, 12 weeks, 24 weeks, 52 weeks, 18 months, and 24 months post-treatment
  Measured using the International Hip Outcome Tool (IHOT12). 12-item self-reported questionnaire assessing function of hip on a scale of 0 to 10, with higher outcomes indicating worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Krych, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No